CLINICAL TRIAL: NCT01865461
Title: Evaluation of MRI Sequences in Hepatic Overload.
Acronym: HEPAT_MR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00197-38
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2020-03

CONDITIONS: Iron and Fat Hepatic Overload
Keywords: Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
MRI, without any contrast injection, allows a non-invasive evaluation and quantification of hepatic overloads, especially iron (liver iron content LIC) and fat (steatosis) overloads, but in certain clinical circumstances, cases require to improve performances. The aim of the study is to add to MRI scans which currently must be performed innovative sequences appropriate for the clinical question to overall appreciate on a varied range of patients their quality, their robustness, their relative performance and, for patients having a biopsy, their accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Patients with or suspected clinically to be with a hepatic overload pathology (hepatic iron and/or fat overload) and who need a diagnostic or pre-therapeutic MRI from his initial management or during his monitoring,
* Patient able to provide written informed consent and can understand and comply with the requirements of the study
* Patient having received the information about the protocol and having not expressed his opposition to participate.

Exclusion Criteria:

Due to MRI :

* pacemaker or defibrillator,
* MRI non-compatible heart valve,
* clips, stents, coils, etc… non-compatible with MRI,
* cochlear implants,
* neuronal or peripheric simulator,
* intra-orbital or encephalic metallic foreign body, foreign body close to eyes, foreign body near the eyes, injury by metallic luster (war, ball),
* endoprosthesis received since less than 4weeks and osteosynthesis equipment received since less than 6 weeks,
* claustrophobia,
* pump, tattoo, permanent make-up, intrauterine device, patch,
* metal, magnetic, non-removable and in the area of the analyse field material

Other criteria :

* unstable hemodynamic state, acute respiratory insufficiency, hemodynamically unstable acute respiratory failure, poor general condition or the necessity of a continuous monitoring incompatible with the MRI constraint,
* adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty,
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or suspected clinically to be with a hepatic overload pathology (hepatic iron and/or fat overload)
Sampling Method: Non-Probability Sample
Enrollment: 706 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quantification deviations of hepatic iron and fat overloads between the new sequences and the conventional sequences. | 18 months
  Evaluation of the robustness and the relative accuracy, comparison of sequences currently performed in daily clinical practice, of hepatic iron and fat content quantification with non-invasive new abdominal MRI sequences.

SECONDARY OUTCOMES:
Analysis of the accuracy of quantification: of the iron concentration against biochemical, semi-quantitative histological or subtracted iron volume compared to the hepatic volume analysis | 18 months
  Evaluation of the accuracy of these new MRI sequences for hepatic iron and fat quantification, when patients have had in their normal care and management a biopsy or a bleedings subtracted iron volume leading to a desaturation.

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, France